CLINICAL TRIAL: NCT00601406
Title: Radiogenomics: Assessment of Polymorphisms for Predicting the Effects of Radiotherapy (RAPPER)
Brief Title: Study of DNA Mutations in Predicting the Effect of External-Beam Radiation Therapy in Patients With Early Breast Cancer, Localized Prostate Cancer, or Gynecological Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Christie NHS Foundation Trust (Other)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000581139; CHNT-RAPPER; EU-20798
Record Dates: First submitted 2008-01-25; First posted 2008-01-28 (Estimated); Last update posted 2013-08-26 (Estimated); Status verified 2008-04

CONDITIONS: Breast Cancer; Cervical Cancer; Endometrial Cancer; Fallopian Tube Cancer; Ovarian Cancer; Primary Peritoneal Cavity Cancer; Prostate Cancer; Sarcoma; Vaginal Cancer; Vulvar Cancer
Keywords: male breast cancer; stage IA breast cancer; stage IB breast cancer; stage II breast cancer; stage I prostate cancer; stage IIB prostate cancer; stage IIA prostate cancer; stage III prostate cancer; stage IA cervical cancer; stage IB cervical cancer; stage IIA cervical cancer; stage IIB cervical cancer; stage III cervical cancer; stage IVA cervical cancer; stage IVB cervical cancer; stage I vaginal cancer; stage II vaginal cancer; stage III vaginal cancer; stage IVA vaginal cancer; stage IVB vaginal cancer; stage IA vulvar cancer; stage IB vulvar cancer; stage II vulvar cancer; stage IIIC vulvar cancer; stage IIIA vulvar cancer; stage IIIB vulvar cancer; stage IVB vulvar cancer; stage IA ovarian epithelial cancer; stage IB ovarian epithelial cancer; stage IC ovarian epithelial cancer; stage IA ovarian germ cell tumor; stage IB ovarian germ cell tumor; stage IC ovarian germ cell tumor; stage IIA ovarian epithelial cancer; stage IIB ovarian epithelial cancer; stage IIC ovarian epithelial cancer; stage IIA ovarian germ cell tumor; stage IIB ovarian germ cell tumor; stage IIC ovarian germ cell tumor; stage IIIA ovarian epithelial cancer; stage IIIB ovarian epithelial cancer; stage IIIC ovarian epithelial cancer; stage IIIA ovarian germ cell tumor; stage IIIB ovarian germ cell tumor; stage IIIC ovarian germ cell tumor; stage IV ovarian epithelial cancer; stage IV ovarian germ cell tumor; stage II endometrial carcinoma; ovarian stromal cancer; ovarian sarcoma; stage IA fallopian tube cancer; stage IB fallopian tube cancer; stage IC fallopian tube cancer; stage IIA fallopian tube cancer; stage IIB fallopian tube cancer; stage IIC fallopian tube cancer; stage IIIA fallopian tube cancer; stage IIIB fallopian tube cancer; stage IIIC fallopian tube cancer; stage IV fallopian tube cancer; recurrent primary peritoneal cavity cancer; stage IA primary peritoneal cavity cancer; stage IB primary peritoneal cavity cancer; stage IC primary peritoneal cavity cancer; stage IIA primary peritoneal cavity cancer; stage IIB primary peritoneal cavity cancer; stage IIC primary peritoneal cavity cancer; stage IIIA primary peritoneal cavity cancer; stage IIIB primary peritoneal cavity cancer; stage IIIC primary peritoneal cavity cancer; stage IV primary peritoneal cavity cancer; stage IA endometrial carcinoma; stage IB endometrial carcinoma; stage IIIA endometrial carcinoma; stage IIIB endometrial carcinoma; stage IIIC endometrial carcinoma; stage IVA endometrial carcinoma; stage IVB endometrial carcinoma; stage IA uterine sarcoma; stage IB uterine sarcoma; stage IC uterine sarcoma; stage IIA uterine sarcoma; stage IIB uterine sarcoma; stage IIIA uterine sarcoma; stage IIIB uterine sarcoma; stage IIIC uterine sarcoma; stage IVA uterine sarcoma; stage IVB uterine sarcoma
MeSH Terms: conditions — Breast Neoplasms; Uterine Cervical Neoplasms; Endometrial Neoplasms; Fallopian Tube Neoplasms; Ovarian Neoplasms; Prostatic Neoplasms; Sarcoma; Vaginal Neoplasms; Vulvar Neoplasms; Breast Neoplasms, Male; Carcinoma, Ovarian Epithelial | interventions — Gene Expression Profiling; Gene Rearrangement; Amplified Fragment Length Polymorphism Analysis; Radiotherapy

INTERVENTIONS:
Genetic: gene expression analysis
Genetic: gene rearrangement analysis
Genetic: polymorphism analysis
Other: laboratory biomarker analysis
Radiation: radiation therapy

SUMMARY:
RATIONALE: Studying samples of blood from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer. It may also help doctors predict how patients will respond to treatment.

PURPOSE: This clinical trial is evaluating DNA mutations in predicting the effect of external-beam radiation therapy in patients with early breast cancer, localized prostate cancer, or gynecologic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To test the hypothesis that an association between common genetic variations, reported by single nucleotide polymorphisms (SNP) in relevant candidate genes, is associated with individual patient variability in normal tissue radiation response and toxicity.

Secondary

* To compare different clinical scoring systems for late normal tissue effects, specifically Late Effect of Normal Tissue Subjective Objective Management Analysis (LENT SOMA), Radiation Therapy Oncology Group (RTOG), quality of life, and in a subset common terminology criteria (CTC) version 3.
* To compare clinical scoring systems with analytical measures of normal tissue outcome in a minority of patients, using volume change in the breast measured by laser camera.
* To correlate family history information with SNP analysis to produce a polymorphism risk score (PRS) for family history.
* To compare a detailed 3D dose-volume analysis in a subset of patients with late effects and SNP results.
* To correlate actuarial analysis of late effects changes over time with PRS.
* To conduct PRS analyses against tumor control probability (TCP), using survival as a surrogate for TCP where necessary, and normal tissue complications vs tumor control probability.

OUTLINE: This is a multicenter study.

Patients are recruited from clinical trials in which their late normal tissue effects have been measured. Blood samples are collected from these patients for analysis of genetic variation by DNA extraction and single nucleotide polymorphism analysis. Sixty different genes, including those involved in cell cycle checkpoint control, DNA damage recognition and repair, induction of apoptosis, and cytokine production (including TGFβ pathways) are assessed.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Patients must have received curative external-beam radiotherapy within the context of a formal clinical study for any of the following:

  * Early breast cancer after breast-conserving surgery
  * Localized prostate cancer
  * Gynecological cancer (may have also received brachytherapy)
* Venous blood samples must be available
* Patients will be identified from the following clinical studies:

  * Cambridge intensity-modulated radiotherapy breast randomized trial
  * RT01 prostate radiotherapy randomized trial/other prostate trials
  * Christie hospital breast, prostate, and gynecological cancer radiotherapy patients
* Must have minimum follow up with late normal tissue effect scoring for two years available

PATIENT CHARACTERISTICS:

* No other malignancy prior to treatment for the specified tumor types except basal cell or squamous cell carcinoma of the skin or in situ carcinoma

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2200 (Estimated)
Dates: Start 2006-03; Primary Completion 2008-02 (Estimated)

PRIMARY OUTCOMES:
Correlation of association between common genetic variations, reported by single nucleotide polymorphisms (SNP) in relevant candidate genes, with individual patient variability in normal tissue radiation response and toxicity

SECONDARY OUTCOMES:
Comparison of different clinical scoring systems for late normal tissue effects
Comparison of clinical scoring systems with analytical measures of normal tissue outcome using volume change in the breast measured by laser camera
Correlation of family history information with SNP analysis to produce a polymorphism risk score (PRS)
Comparison of detailed 3D dose-volume analysis with late effects and SNP results
Correlation of actuarial analysis of late effects changes over time with PRS
PRS analyses against tumor control probability (TCP), using survival as a surrogate for TCP where necessary, and normal tissue complications vs tumor control probability

CONTACTS AND LOCATIONS:
Overall Officials: Catherine West, Study Chair — The Christie NHS Foundation Trust
Locations (11):
- United Kingdom (11):
  - Sussex Cancer Centre at Royal Sussex County Hospital, Brighton, England
  - Bristol Haematology and Oncology Centre, Bristol, England
  - Addenbrooke's Hospital, Cambridge, England
  - Ipswich Hospital, Ipswich, England
  - Christie Hospital, Manchester, England
  - Clatterbridge Centre for Oncology, Merseyside, England
  - Whiston Hospital, Prescot, England
  - Cancer Research Centre at Weston Park Hospital, Sheffield, England
  - Southport and Formby District General Hospital, Southport, England
  - Royal Marsden - Surrey, Sutton, England
  - Warrington Hospital NHS Trust, Warrington, England